CLINICAL TRIAL: NCT05134415
Title: A Randomized, Single-Blind, Two-Arm, Cross-Over Study to Compare Use of Two Tobacco and Two Menthol Flavor e-Liquids in Electronic Nicotine Delivery System Users
Brief Title: Use Behavior, Nicotine Uptake, and Subjective Effects Comparison of Tobacco and Menthol e-Liquids by ENDS Consumers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cheerain HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: RELX-004
Record Dates: First submitted 2021-11-13; First posted 2021-11-26 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Electronic Cigarette Use
Keywords: Electronic Nicotine Delivery System; Nicotine; Topography; Pharmacokinetics; E-cigarette; Subjective effects
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to the specific tobacco or menthol flavor variant used during each study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Product Use Sequence 1 (Experimental): Period 1 - RELX ENDS tobacco flavor 1 Period 2 - RELX ENDS tobacco flavor 2
  Interventions: Other: RELX ENDS Tobacco Flavor 1; Other: RELX ENDS Tobacco Flavor 2
- Product Use Sequence 2 (Experimental): Period 1 - RELX ENDS tobacco flavor 2 Period 2 - RELX ENDS tobacco flavor 1
  Interventions: Other: RELX ENDS Tobacco Flavor 1; Other: RELX ENDS Tobacco Flavor 2
- Product Use Sequence 3 (Experimental): Period 1 - RELX ENDS menthol flavor 1 Period 2 - RELX ENDS menthol flavor 2
  Interventions: Other: RELX ENDS Menthol Flavor 1; Other: RELX ENDS Menthol Flavor 2
- Product Use Sequence 4 (Experimental): Period 1 - RELX ENDS menthol flavor 2 Period 2 - RELX ENDS menthol flavor 1
  Interventions: Other: RELX ENDS Menthol Flavor 1; Other: RELX ENDS Menthol Flavor 2

INTERVENTIONS:
Other: RELX ENDS Tobacco Flavor 1 — 2-week ad libitum use of the RELX ENDS tobacco flavor 1
  Arms: Product Use Sequence 1; Product Use Sequence 2
Other: RELX ENDS Tobacco Flavor 2 — 2-week ad libitum use of the RELX ENDS tobacco flavor 2
  Arms: Product Use Sequence 1; Product Use Sequence 2
Other: RELX ENDS Menthol Flavor 1 — 2-week ad libitum use of the RELX ENDS menthol flavor 1
  Arms: Product Use Sequence 3; Product Use Sequence 4
Other: RELX ENDS Menthol Flavor 2 — 2-week ad libitum use of the RELX ENDS menthol flavor 2
  Arms: Product Use Sequence 3; Product Use Sequence 4

SUMMARY:
This study is being conducted to evaluate the impact of within-flavor category (tobacco and menthol) differences in e-liquid flavors on product use behaviors, nicotine uptake, and subjective effects by current ENDS consumers when used in a closed-system electronic nicotine delivery system (ENDS).

ELIGIBILITY:
Inclusion Criteria:

1. Is 22 to 65 years of age, inclusive, at the time of consent.
2. Has used a closed-system ENDS product on most days during the 60 days prior to Screening (no use on up to 8 days total is allowed). Dual use with open-system products will be allowed provided that the closed-system is the predominant system used (based on self-reported volume of e-liquid used).
3. Reports a tobacco or menthol/mint flavored e-liquid as the most commonly used flavor (based on self-reported volume of e-liquid used) during the 30 days prior to screening.
4. Agrees to maintain product use described in Criteria 3 and 4 from Screening through Test Visit 1.
5. Has a urine cotinine concentration ≥ 200 ng/mL at Screening.
6. Has an ECO concentration < 10 ppm at Screening and Test Visit 1.
7. If female, must meet one of the following criteria:

   If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to the first product use and during the study. An acceptable method of contraception includes one of the following:
   * Abstinence from heterosexual intercourse
   * Hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
   * Intrauterine device (with or without hormones) OR agrees to use a double barrier method (e.g., condom and spermicide) during the study.

   If a female of non-childbearing potential - should be surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion) or in a menopausal state (at least 1 year without menses).
8. Is willing to comply with the requirements of the study.
9. Provides voluntary consent to participate in the study as documented on the signed ICF.

Exclusion Criteria:

1. Has a history or presence of clinically significant uncontrolled gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that would jeopardize the safety of the subject or impact the validity of the study results.
2. Has a clinically significant abnormal finding on the physical examination, medical history, vital signs, ECG, or clinical laboratory results at Screening, including, but not limited to, the following:

   1. Has a history of drug or alcohol abuse within 12 months of Screening.
   2. Has a systolic BP <90 mmHg or >160 mmHg, diastolic BP <40 mmHg or >95 mmHg, or HR <40 bpm or >99 bpm at Screening.
   3. Has previously been diagnosed with any form of cancer, except for basal cell or squamous epithelial carcinomas of the skin that have been resected.
   4. Has been treated chronically for depression, diabetes, asthma, emphysema, or chronic obstructive pulmonary disease within 12 months of Test Visit 1.
3. Has had an acute illness (e.g., upper respiratory infection, viral infection) within 14 days prior to Test Visit 1 that would jeopardize the safety of the subject or impact the validity of the study results.
4. Subjects who, in the judgment of the study physician, have recent or active COVID 19 infection, as evidenced by the following:

   1. Endorsement of symptoms that could indicate COVID-19 during screening and/or
   2. Body temperature ≥100.4°F and/or
   3. Laboratory test results suggestive of active or recent exposure to SARS CoV 2.
5. Has a BMI greater than 40.0 kg/m2 or less than 18.0 kg/m2 at Screening.
6. Is allergic to or intolerant of components of the product e-liquid, including but not limited to, menthol, propylene glycol, or glycerin.
7. Has a positive urine drug or alcohol test at Screening..
8. If female, has a positive pregnancy test, is breastfeeding or lactating, or intends to become pregnant from Screening through Test Visit 3.
9. Is a current combustible cigarette, cigar, or little cigar smoker at Screening (more than 5 product uses in the previous 30 days).
10. Has used other tobacco- or nicotine-containing products other than ENDS products (e.g., combustible cigarettes, cigars, or little cigars, snuff, pouches, chewing tobacco, nicotine inhalers, nicotine patches, nicotine sprays, nicotine lozenges, or nicotine gum) from 14 days prior to Test Visit 1.
11. Has used any products for the purpose of smoking/vaping cessation, including, but not limited to, nicotine replacement therapies, varenicline (Chantix), or bupropion (Zyban) from 30 days prior to Screening through Test Visit 3.
12. Draws aerosol from the usual brand ENDS into the mouth and throat but does not inhale as observed by the clinic staff during Screening.
13. Is postponing a planned vaping quit attempt in order to participate in the study.
14. Has donated plasma within 7 days prior to Test Visit 1.
15. Has provided a whole blood donation, had significant blood loss, or received whole blood or a blood product transfusion within 56 days prior to Test Visit 1.
16. Has participated in a previous clinical study for a tobacco product or an investigational drug, device, or biologic, within 30 days or 5 times the half-life of the product (whichever is longer) prior to Test Visit 1.
17. Is or has a first-degree relative (e.g., spouse, parent, sibling, child) who is a current or former employee of a tobacco or ENDS manufacturer (including the Sponsor) or is a named party or class representative in litigation with the tobacco or ENDS industry.
18. Is or has a first-degree relative (e.g., spouse, parent, sibling, child) who is a current employee of the clinic site(s).
19. Has previously been withdrawn from or has completed this study.
20. In the opinion of an Investigator, the subject should not participate in this study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Study product use - daily pod use | 14 days
  The number of pods used per day during the 14-day ambulatory period

SECONDARY OUTCOMES:
Study product use - e-liquid consumption per pod | 14 days
  The amount of e-liquid consumed per pod during the 14-day ambulatory period
Study product use - e-liquid consumption per day | 14 days
  The amount of e-liquid consumed each day during the 14-day ambulatory period
Puff topography - number of puffs | 5 minutes
  Number of puffs taken from the study products during the PK Session
Puff topography - duration of puffs | 5 minutes
  Duration of puffs taken from the study products during the PK Session
Puff topography - volume of puffs | 5 minutes
  Volume of puffs taken from the study products during the PK Session
Puff topography - peak flow rate of puffs | 5 minutes
  Peak flow rate of puffs taken from the study products during the PK Session
Puff topography - average flow rate of puffs | 5 minutes
  Average flow rate of puffs taken from the study products during the PK Session
Puff topography - inter-puff interval | 5 minutes
  Inter-puff interval of puffs taken from the study products during the PK Session
Study product use - e-liquid consumption (PK session) | 5 minutes
  Change in pod weight of pods used during the PK Session
Subjective effects - dependence | 14 days
  Nicotine dependence as measured by the Penn State Electronic Cigarette Dependence Index (PSECDI) total score. Total scores may range from 0 to 20, with higher levels of dependence associated with higher scores.
Subjective effects - craving | 14 days
  Craving as measured by the Questionnaire of Vaping Craving (QVC) average score. Questionnaire responses are measured on a Likert scale range of 1 [strongly disagree] to 7 [strongly agree].
Subjective effects - withdrawal symptoms | 14 days
  Withdrawal symptoms as measured by the Minnesota Tobacco Withdrawal Scale - Revised (MTWS-R), which includes the DSM-5 and craving items from the MTWS. Questionnaire responses are measured on a Likert scale range of 0 [none] to 4 [severe]).
Subjective effects - product effects | 14 days
  Product effects as measured by the Modified Product Evaluation Scale (mPES) satisfaction, psychological reward, aversion, and relief subscale and individual item scores. Questionnaire responses are measured on a Likert scale range of 1 [not at all] to 7 [extremely].
Subjective effects - future intent to use product | 14 days
  Future intent to use the product as measured by the Future Intent to Use Questionnaire (FIU). Questionnaire responses are measured on a Likert scale range of 1 [extremely unlikely] to 7 [extremely likely].
Subjective effects - maximum acute urge to vape reduction | 30 minutes
  Maximum urge to vape reduction (Emax_R) as measured by responses to the Urge to Vape questionnaire (visual analog scale range of "Not at All" to "Extreme")
Subjective effects - overall acute urge to vape reduction | 30 minutes
  Overall urge to vape reduction (AOEC0-30) as measured by responses to the Urge to Vape questionnaire (visual analog scale range of "Not at All" to "Extreme")
Subjective effects - time to maximum acute urge to vape reduction | 30 minutes
  Time to the maximum urge to vape reduction (TEmax_R) as measured by responses to the Urge to Vape questionnaire (visual analog scale range of "Not at All" to "Extreme")
Nicotine uptake - maximum nicotine concentration | 30 minutes
  Baseline-adjusted maximum plasma nicotine concentration [Cmax]
Nicotine uptake - overall nicotine uptake | 30 minutes
  Baseline-adjusted area under the nicotine concentration-time curve [AUC(0-30)]
Nicotine uptake - time to maximum nicotine concentration | 30 minutes
  Time of the maximum post-baseline nicotine concentration [Tmax]
Safety and tolerability - adverse events | 14 days
  Incidence of product-use emergent adverse events
Safety and tolerability - product malfunction or misuse | 14 days
  Incidence of product malfunction or misuse

CONTACTS AND LOCATIONS:
Overall Officials: Donald Graff, PharmD, Study Director — RELX International
Locations (1):
- Los Angeles Clinical Trials, Burbank, California, United States

IPD SHARING:
Plan to Share IPD: No